CLINICAL TRIAL: NCT00410657
Title: A Phase II Study to Evaluate Low-Dose Alemtuzumab as a Glucocorticoid-Sparing Agent for Initial Systemic Treatment of Acute Graft-Versus-Host Disease
Brief Title: Alemtuzumab and Glucocorticoids in Treating Newly Diagnosed Acute Graft-Versus-Host Disease in Patients Who Have Undergone a Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: 2096.00; FHCRC-2096.00; CDR0000523371 (Registry Identifier: PDQ)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: graft versus host disease; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; splenic marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; aggressive, noncontiguous stage II adult non-Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood myelodysplastic syndromes
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Carcinoma, Ovarian Epithelial; Aggression; Hodgkin Disease; Testicular Neoplasms | interventions — Alemtuzumab; Methylprednisolone; Prednisone; Flow Cytometry; Immunologic Techniques

INTERVENTIONS:
Biological: alemtuzumab
Drug: methylprednisolone
Drug: prednisone
Other: flow cytometry
Other: immunologic technique
Other: pharmacological study

SUMMARY:
RATIONALE: Alemtuzumab and glucocorticoids, such as prednisone or methylprednisolone, may be an effective treatment for acute graft-versus-host disease caused by a donor stem cell transplant.

PURPOSE: This phase II trial is studying how well giving alemtuzumab together with glucocorticoids works in treating newly diagnosed acute graft-versus-host disease in patients who have undergone donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the administration of low-dose alemtuzumab at the onset of acute graft-versus-host disease can accelerate withdrawal of glucocorticoids and decrease nonrelapsing mortality in patients who have undergone myeloablative allogeneic stem cell transplantation.

OUTLINE: This is an open-label, nonrandomized study.

Within 72 hours of beginning glucocorticoid therapy, patients receive alemtuzumab IV over at least 2 hours on days 1 and 2. If graft-versus-host disease (GVHD) responds well during days 1-14 but returns between days 28 and 56, patients are eligible to receive 2 additional doses of alemtuzumab.

Patients receive glucocorticoid therapy comprising methylprednisolone IV or oral prednisone daily until objective evidence of improvement in manifestations of GVHD. Patients with resolved or significantly improved GVHD receive treatment until day 10 followed by an accelerated taper until day 72 if no flare up of GVHD occurs during the glucocorticoid taper. Patients with recurrent or progressive GVHD during the accelerated taper are treated for 5-7 days before resuming a less rapid taper. Patients with no improvement may receive secondary therapy with alternative immunosuppressive medications at the discretion of the managing physician. Treatment continues in the absence of progressive GVHD of at least 3 days duration during days 2-10; persisting GVHD without improvement between days 10-14; recurrent or progressive GVHD after day 10 that does not respond within 3 days to topical immunosuppressive therapy; and/or an increase in the systemic glucocorticoid dose by two taper steps; or unacceptable toxicity.

Patients undergo blood collection at baseline and then periodically during study treatment for pharmacokinetics and quantification of viral loads for human herpes virus 6, adenovirus, Epstein-Barr virus, and cytomegalovirus. Samples are also examined by flow cytometry for B- and T-cell quantification at baseline, periodically during study treatment, and at 1 year after transplantation.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 53 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute graft-versus-host disease (GVHD)

  * Grade IIB-IV disease
* Requires glucocorticoids for treatment of GVHD, as indicated by 1 of the following:

  * Initial treatment with prednisone or methylprednisolone at 2 mg/kg is indicated (in the judgement of the attending physician) by any of the following:

    * Severity of GVHD requires hospitalization
    * GVHD manifestations include symptoms other than anorexia, nausea, and vomiting
    * GVHD begins within 2-3 weeks after hematopoietic stem cell transplantation (HSCT)
    * GVHD manifestations progress rapidly from 1 day to the next before treatment
  * Initial treatment with prednisone or methylprednisolone at 1 mg/kg did not produce adequate clinical improvement within the first 4 days (in the judgement of the attending physician)
* Has undergone allogeneic HSCT with myeloablative conditioning

  * No nonmyeloablative conditioning or autologous HSCT
* No primary treatment of acute GVHD with methylprednisolone at any of the following doses:

  * More than 2 mg/kg/day at any time
  * 2 mg/kg/day for > 72 hours
  * 1 mg/kg/day for > 96 hours
* No presence of distinctive or diagnostic manifestations of chronic GVHD
* No relapsed, refractory, or secondary malignancy

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 20-100% OR Lanksy PS 20-100%
* Life expectancy ≥ 1 month
* Absolute neutrophil count ≥ 500/mm^3
* Negative pregnancy test
* No Mini Mental State Exam score < 24/30 or confusion (for patients > 12 years of age)
* No history of type I hypersensitivity reaction to alemtuzumab or any of its components
* No increasing levels of viremia by serial quantitative viral plasma polymerase chain reaction assays
* No invasive viral or fungal disease that does not respond to appropriate antiviral or antifungal medications

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No systemic immunosuppression tapered or stopped for treatment of leukemic relapse or minimal residual disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2006-07; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with methylprednisolone (MP)-equivalent glucocorticoid doses ≤ 0.75 mg/kg on day 28 after starting therapy for graft-versus-host disease (GVHD)

SECONDARY OUTCOMES:
Total cumulative dose of MP-equivalent treatment during the first 8 weeks after study entry
Proportion of patients with complete response, measured weekly through day 56
Incidence of secondary systemic therapy for acute GVHD
Cumulative acute GVHD activity index score at day 56
Incidence of chronic GVHD at 1 year
Nonrelapsing mortality at 1 year
Survival at 1 year
Cumulative incidence of opportunistic infections at 1 year
Cumulative incidence of recurrent or progressive malignancy at 1 year
Peripheral blood CD4, CD8, CD19, and CD16/56 counts at baseline and then periodically for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Carpenter, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States